CLINICAL TRIAL: NCT01573312
Title: A Randomized, Double-Blinded, Controlled, Phase I Study in Healthy Adults to Assess the Safety, Reactogenicity, and Immunogenicity of Intramuscular Subvirion Inactivated Monovalent Influenza A/H5N1 Virus Vaccine Administered With and Without AS03 Adjuvant: Standard & Systems Biology Analyses
Brief Title: H5N1 Vaccination With and Without AS03: Systems Biology Analysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-0074; N01AI80007C; VTEU 02-2011
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2013-07

CONDITIONS: Influenza
Keywords: influenza, vaccine, H5N1, monovalent, adjuvant, ASO3
MeSH Terms: conditions — Influenza, Human; Influenza in Birds | interventions — AS03 adjuvant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Inactivated monovalent influenza A/H5N1 with ASO3 adjuvant (Experimental): Ten subjects will be vaccinated with 3.75 micrograms(mcg) of H5N1 hemagglutinin plus AS03 given intramuscularly in two doses 28 days apart.
  Interventions: Drug: ASO3 Adjuvant; Biological: Influenza A/H5N1 Vaccine
- Inactivated monovalent influenza A/H5N1 without ASO3 adjuvant (Experimental): Ten subjects will be vaccinated with 3.75 mcg of H5N1 hemagglutinin alone, given intramuscularly, in two doses 28 days apart.
  Interventions: Biological: Influenza A/H5N1 Vaccine

INTERVENTIONS:
Drug: ASO3 Adjuvant — 3.75 mcg of H5N1 hemagglutinin plus AS03, will be administered in 2 doses 28 days apart.
  Arms: Inactivated monovalent influenza A/H5N1 with ASO3 adjuvant
Biological: Influenza A/H5N1 Vaccine — 3.75 mcg of H5N1 hemagglutinin plus AS03 or 3.75 mcg of H5N1 hemagglutinin alone will be administered in two doses 28 days apart.

SUMMARY:
This is a single center, randomized, double-blinded, controlled, Phase I, small targeted prospective study in healthy male and non-pregnant female subjects, 18 to 49 years old, inclusive, designed to determine the safety, reactogenicity, and immunogenicity of an intramuscular subvirion inactivated monovalent influenza A/H5N1 (HA of A/Indonesia/05/2005) virus vaccine manufactured by Sanofi Pasteur administered at 3.75 mcg per dose given with or without AS03 adjuvant manufactured by GSK. In the study, each subject will receive two doses administered 28 days apart. This study will use a systems biology approach to assess the human early gene and protein signatures expressed at Days 1, 3, 7, and 28 after the first vaccination. The systems data will be integrated with immunogenicity and reactogenicity data to develop a systems model of the human immune response to A/H5N1 vaccine with or without AS03 adjuvant.

DETAILED DESCRIPTION:
The long term goals of this project are to identify RNA or protein biomarkers within 1 to 7 days after vaccination in peripheral blood that will predict a successful immune response and protection against disease. Adjuvants are used to boost the response of vaccines by stimulating the innate immune response. However, the exact mechanism and safety of adjuvants is still debated. Systems biology is the study of complex biological processes as integrated systems with many interacting components. The goal of systems biology is to make biology more predictive. This proposal will use a systems biology approach to identify successful immunization biomarkers. The study will use fresh blood samples and patient data collected in the proposed VTEU-funded study. At selected time points, volunteers' blood samples will be collected and immediately processed. Using these specimens, we will identify and quantify changes in the whole transcriptome and proteome of the major immune cells to identify and quantify changes in gene expression. We will integrate the changes in gene expression with the changes in the immune cells response. We will use mathematical modeling of the accumulated data to identify RNA or protein biomarkers that significantly correlate with the observed serum hemagglutination inhibition assay (HAI) response,cytokine/chemokine response, and cell mediated immunity (CMI) responses. Ultimately, the predictive biomarkers will be the foundation for a simple, rapid, inexpensive test to quickly show protection against a pathogen or foreign agent after vaccination. This is a single center, randomized, double-blinded, controlled, Phase I, small targeted prospective study in healthy male and non-pregnant female subjects, 18 to 49 years old, inclusive, designed to determine the safety, reactogenicity, and immunogenicity of an intramuscular subvirion inactivated monovalent influenza A/H5N1 (HA of A/Indonesia/05/2005) virus vaccine manufactured by Sanofi Pasteur administered at 3.75 mcg per dose given with or without AS03 adjuvant manufactured by GSK. In the study, each subject will receive two doses administered 28 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Are males or non-pregnant females between the ages of 18 and 49 years, inclusive.
* Women of childbearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for >/= 1 year) must agree to practice adequate contraception (that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms or diaphragms with spermicide or foam, intrauterine devices, and licensed hormonal methods) during the study for at least 30 days following the last vaccination. Method of contraception will be captured on the appropriate case report form (CRF).
* Are in good health, as determined by vital signs (oral temperature, pulse and blood pressure), medical history and complete physical examination (without genital and rectal exam) to ensure no existing chronic medical diagnoses or conditions are present.
* For women of childbearing potential, negative urine or serum pregnancy test within 24 hours prior to vaccination.
* Are able to understand and comply with planned study procedures.
* Provide written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Have a known allergy to eggs or other components of the vaccine (including gelatin, formaldehyde, octoxinol-9, thimerosal and chicken protein), or allergy to squalene-based adjuvants.
* Women who are breastfeeding or plan to breastfeed at any given time from the first vaccination until 30 days after the last vaccination.
* Have long term use (defined as taken for 2 weeks or more in total at any time during the past 2 months) of high dose oral or parenteral glucocorticoids (high dose defined as prednisone >/= 20 mg total daily dose, or equivalent dose of other glucocorticoids); or high-dose inhaled steroids (high dose defined as >800 mcg/day of beclomethasone dipropionate or equivalent); or systemic corticosteroids of any dose within the past 4 weeks.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have a diagnosis of schizophrenia, bipolar disease, or other major psychiatric diagnosis.
* Hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
* Receiving systemic, prescription medications for the treatment of chronic medical conditions, unless such use is on a PRN (as needed) basis only. Non-PRN use of systemic, over-the-counter medications and PRN systemic, prescription medication may be allowed if, in the opinion of the investigator, they pose no additional risk to subject safety or assessment of immunogenicity/reactogenicity. Note: Topical, nasal, and inhaled medications; vitamins; and contraceptives are also permitted.
* Received pre-medication with analgesic or antipyretic agents in the 6 hours prior to first vaccination, or planned medication with analgesic or antipyretic in the week following first vaccination. This criterion should not preclude subjects receiving such medication if the need arises. However, pre-medication is to be discouraged.
* Received immunoglobulin or other blood products (with exception of Rho D immune globulin) within the 3 months prior to the first vaccination.
* Received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to the first vaccination or plan receipt of such vaccines within 56 days following the first vaccination. This is inclusive of licensed seasonal influenza vaccines.
* Have an acute or chronic medical condition that, in the opinion of the site principal investigator or appropriate sub-investigator, would render vaccination unsafe, would interfere with the evaluation of responses or is not generally seen in "normal, healthy subjects".
* Have a history of severe reactions following previous immunization with contemporary influenza virus vaccines.
* Have an acute illness, including an oral temperature greater than or equal to 100.4 degree F, within 3 days prior to the first vaccination.
* Pulse is less than 55 bpm or greater than 100 bpm.
* Systolic blood pressure is less than 90 mm Hg or greater than 140 mm Hg.
* Diastolic blood pressure is less than 60 mm Hg or greater than 90 mmHg.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to the first vaccination or expects to receive an experimental agent, other than from participation in this study, during the 14-month study period.
* Are participating or plan to participate in another clinical trial with a licensed product during the 14-month study period.
* Have any condition that, in the opinion of the site principal investigator or appropriate sub-investigator, would place the subject at an unacceptable risk of injury, or render them unable to meet the requirements of the protocol, or confound the interpretation of results.
* Participated in an influenza A/H5 vaccine study in the past in a group receiving vaccine (does not apply to documented placebo recipients) or have a history of A/H5 infection prior to enrollment.
* Have known active HIV, Hepatitis B, or Hepatitis C infection.
* Have a history of alcohol or drug abuse in the last 5 years.
* Plan to travel outside the U.S. in the time between the first vaccination and 56 days following the first vaccination.
* Have a history of Guillain-Barré Syndrome.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05-24 (Actual); Primary Completion 2014-01-02 (Actual); Study Completion 2014-01-02 (Actual)

PRIMARY OUTCOMES:
GMT of neutralizing antibody, proportion of subjects achieving a serum neutralizing antibody titer of 1:40 or greater, and frequency of 4-fold or greater increases of neutralizing antibodies in each group against the subvirion inactivated A/H5N1 virus | Approximately Days:1, 3, 7 and 28, after receipt of the first dose of vaccine.
Occurrence of vaccine associated serious adverse events (SAEs) from the time of first vaccination through 13 months after the first vaccination. | Day 0 through 13 months after receipt of the first dose of vaccine.
Occurrence of solicited local and systemic reactogenicity in the 8 days (Days 0 through Day 7) after each vaccination. | Day 0 through Day 7 after each dose of vaccine
Geometric mean titer (GMT) of the hemagglutination inhibition assay (HAI) antibody, proportion of subjects achieving serum HAI antibody titer 1:40 or greater, & frequency of 4-fold or greater increases of HAI antibodies in each group against the vaccine. | Approximate Days: 1, 3, 7 and 28 after receipt of the first dose of vaccine

SECONDARY OUTCOMES:
GMT of neutralizing antibody, proportion of subjects achieving a serum neutralizing antibody titer of 1:40 or greater, and frequency of 4-fold or greater increases of neutralizing antibodies in each group against the subvirion inactivated A/H5N1 virus | 28 days after receipt of the second dose of vaccine (approximately Day 56).
GMT of HAI antibody, proportion of subjects achieving a serum HAI antibody titer of 1:40 or greater, and frequency of 4-fold or greater increases of HAI antibodies in each group against the subvirion inactivated A/H5N1 virus vaccine | 28 days after receipt of the second dose of vaccine (approximately Day 56).

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Howard LM, Jensen TL, Goll JB, Gelber CE, Bradley MD, Sherrod SD, Hoek KL, Yoder S, Jimenez-Truque N, Edwards K, Creech CB. Metabolomic Signatures Differentiate Immune Responses in Avian Influenza Vaccine Recipients. J Infect Dis. 2024 Sep 23;230(3):716-725. doi: 10.1093/infdis/jiad611. PMID 38181048
- [Derived] Howard LM, Hoek KL, Goll JB, Samir P, Galassie A, Allos TM, Niu X, Gordy LE, Creech CB, Prasad N, Jensen TL, Hill H, Levy SE, Joyce S, Link AJ, Edwards KM. Cell-Based Systems Biology Analysis of Human AS03-Adjuvanted H5N1 Avian Influenza Vaccine Responses: A Phase I Randomized Controlled Trial. PLoS One. 2017 Jan 18;12(1):e0167488. doi: 10.1371/journal.pone.0167488. eCollection 2017. PMID 28099485